CLINICAL TRIAL: NCT01140269
Title: Rapid, Quantitative, PCR-Based Detection Of Staphylococcus Aureus in Burn Sepsis Patients
Brief Title: Rapid Detection of Staphylococcus Aureus in Burn Patients
Acronym: PCR-Staph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Burn Association (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ABA-MCTG-0002
Record Dates: First submitted 2010-06-04; First posted 2010-06-09 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Burns; Sepsis
Keywords: Burn; Sepsis; Infection
MeSH Terms: conditions — Burns; Sepsis; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No PCR testing (No Intervention): Control patients will not have PCR testing. This group will have routine testing and treatment as defined by the standard of care.
- PCR testing (Experimental): PCR will be used in parallel with routine laboratory tests such as culture. Treatment for PCR results will be based on the standard of care. Treatment of the patient will be dependent on the physician's clinical judgment based on existing clinical information including PCR, microbiology, patient physical presentation, and other laboratory results.
  Interventions: Other: PCR test

INTERVENTIONS:
Other: PCR test — PCR samples will test for Staphylococcus aureus (including MRSA) from wound swab and positive blood culture samples to augment treatment decisions. Serial PCR testing will follow after positive results to catalog pathogen loads over the course of treatment in a blinded fashion.
  Arms: PCR testing

SUMMARY:
The purpose of this study is to determine if rapid early detection of the bacteria causing sepsis in burn patients improves patient outcomes.

DETAILED DESCRIPTION:
Burn patients have lost their primary barrier to microorganism invasion and therefore are continually and chronically exposed to pathogens. Ninety-seven percent of patients with >20% total body surface area (TBSA) burns develop septicemia; predominantly involving gram positive cocci including MRSA and methicillin sensitive Staphylococcus aureus. Blood culture (BC) is the traditional detection method for septicemia. However, antibiotics and inadequate sample volumes can impair detection by BC and results can take 3-4 days.

Polymerase chain reaction (PCR) represents a potential adjunct to BC. Pathogens are detected in a growth-independent manner by targeting their genetic make-up. Quantitative determining of pathogen DNA using PCR could aid in determining antimicrobial drug therapy efficacy by providing results on the same testing day as opposed to 3-4 days with BC. PCR may also detect persistent infections during antimicrobial therapy when culture samples are inhibited.

The aims of this study are:(1)to correlate quantitative PCR results with that of the BC; (2) to test the clinical application of PCR results with clinical outcomes of treatment of presumptive diagnosis of staphylococcal sepsis.

ELIGIBILITY:
Inclusion Criteria:

* 20% or > TBSA burns at hospital admission
* will require BC during hospital stay
* Patient/surrogate able to sign consent

Exclusion Criteria:

* allergic to nafcillin, cefazolin, vancomycin, linezolid, and/or daptomycin
* on antibiotic(s) prior to first BC

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2010-05-30 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Correlation of PCR results with blood culture results | 72 hours after positive blood culture results

SECONDARY OUTCOMES:
Duration of signs of infection | 14 days after the administrationof anti-Staphylococcus therapy
Duration of antibiotic use | 14 days after administration of antimicrobial therapy
Correlation of PCR result with mortality | Day 28 of intensive care unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Nam Tran, PhD, Principal Investigator — University of California, Davis
Locations (4):
- United States (4):
  - University of California Davis Medical Center-Regional Burn Center, Sacramento, California
  - University of Miami Health System, Miami, Florida
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Harborview Medical Center, Seattle, Washington